CLINICAL TRIAL: NCT06987318
Title: A Phase I Study to Evaluate the Safety and Antiviral Activity of Two Human Monoclonal Antibodies (VRC07-523LS and PGT121.414.LS) During Analytic Treatment Interruption in Participants Living With HIV Who Initiated ART During Acute/Early HIV-1 Infection
Brief Title: A Study to Evaluate the Safety and Antiviral Activity of Two Human Monoclonal Antibodies (VRC07-523LS and PGT121.414.LS) During Analytic Treatment Interruption in Participants Living With HIV Who Initiated ART During Acute/Early HIV-1 Infection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Monogram Biosciences (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A5389
Record Dates: First submitted 2025-04-25; First posted 2025-05-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection
Keywords: Suppressive Antiretroviral Therapy; Acute HIV-1; Broadly neutralizing antibody; Antibodies; HIV; HIV antibody; HIV Broadly neutralizing antibody

STUDY DESIGN:
Intervention Model Description: Enrollment will be opened to Arm A first. Once Arm A enrollment is completed, enrollment to Arm B will be opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Biological: VRC07-523LS; Biological: PGT121.414.LS
- Arm B (Experimental)
  Interventions: Biological: VRC07-523LS; Biological: PGT121.414.LS

INTERVENTIONS:
Biological: VRC07-523LS — Administered by Intravenous (IV) infusion at Week 0 and 12 weeks later
Biological: PGT121.414.LS — Administered by IV infusion at Week 0

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of combination broadly neutralizing antibodies (bNAbs), to induce HIV-1 control during analytic treatment interruption (ATI).

DETAILED DESCRIPTION:
This study is an open-label, two-arm, multi-step phase I study evaluating a combination of two broadly neutralizing antibodies (bNAbs), VRC07-523LS and PGT121.414.LS, in people living with HIV (PWH) who started antiretroviral therapy (ART) during acute/early infection. Participants will receive PGT121.414.LS and VRC07-523LS prior to undergoing an analytical treatment interruption (ATI). Participants will restart ART and continue follow-up after ATI to confirm viral suppression.

Participants will be screened for eligibility and have a pre-entry visit. After determination of eligibility, participants will be enrolled sequentially into Arm A (n=20) and then Arm B (n=20). The study consists of three steps including an analytic treatment interruption.

Arm A:

* Step 1: Participants remain on ART and will receive an infusion of VRC07-523LS and PGT121.414.LS at study entry.
* Step 2: Participants will interrupt their ART and receive a second infusion of VRC07-523LS 12 weeks after the initial infusion. Participants will be monitored closely for indications to resume ART.
* Step 3: Upon meeting ART restart criteria in Step 2; participants will resume ART and be followed for up to 24 weeks.

Arm B:

* Step 1: Participants remain on ART and will receive an infusion of VRC07-523LS and PGT121.414.LS at study entry and a second infusion of VRC07-523LS 12 weeks later.
* Step 2: Participants will interrupt their ART. Participants will be monitored closely for indications to resume ART.
* Step 3: Upon meeting ART restart criteria in Step 2; participants will resume ART and be followed for up to 24 weeks.

Participation in both arms will last up to 98 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness of participant to provide informed consent.
* Initiation of combination ART within 90 days of acute HIV diagnosis as defined by any of the criteria listed below:

  * A negative HIV Ab or HIV Ag/Ab Combination Assay and a detectable HIV-1 RNA (qualitative or quantitative) or a subsequently positive Western blot (WB) or equivalent HIV-1 confirmatory assay (e.g. Geenius assay) if no positive HIV-1 RNA test was available.
  * A positive HIV Ab or HIV Ag/Ab Combination Assay or p24 antigen test and a negative or indeterminate HIV confirmatory/differentiating test with a detectable HIV-1 RNA (qualitative or quantitative).
  * A positive HIV Ab or HIV-1 RNA or p24 antigen and positive WB or Geenius HIV-1/HIV-2 Supplemental Assay that is negative for p31 band.
  * Two different rapid HIV tests with discordant results followed by subsequently positive HIV serum antibody and/or HIV-1 RNA tests.
  * A positive HIV antibody test according to standard criteria obtained within 60 days after an initial negative or indeterminate HIV antibody, antigen, or nucleic acid amplification.
* For women who are able to become pregnant, negative serum or urine pregnancy test within 48 hours prior to Step 1 entry.
* All study candidates must agree not to participate in an assisted conception process (e.g., sperm donation, intrauterine insemination, in vitro fertilization) from the screening visit until 12 weeks after the final study visit.
* Women who can become pregnant and are engaging in sexual activity that could lead to pregnancy must agree to use one highly effective method of contraception from Step 1 entry until 12 weeks after the final study visit.
* Willingness to use barrier protection (male or female) during sexual activity during ATI and through confirmed viral resuppression.
* Weight ≥50 kg and ≤150 kg at screening.
* On stable suppressive ART for at least 12 months prior to Step 1 entry. No known ART interruption for longer than 14 days within 12 months prior to Step 1 entry. No more than two known ART interruptions of a duration between 14 and 60 consecutive days since initiation of ART.
* ART regimens must contain a protease inhibitor (PI) or integrase strand transfer inhibitor (INSTI) as one of the active drugs in the ART regimen at the time of Step 1 entry.
* CD4+ cell count of >450 cells/mL obtained within 60 days prior to Step 1 entry.
* Within 60 days prior to Step 1 entry, plasma HIV-1 RNA < 50 copies/mL of plasma.
* Plasma HIV-1 RNA <50 copies/mL (or below the assay limit of quantification if the local assay limit of quantification is >50 copies/mL) since initial viral suppression on ART and for at least 1 year prior to Step 1 entry.
* Willingness to participate in an ATI.
* The following laboratory values obtained within 60 days prior to Step 1 entry:

  * Absolute neutrophil count (ANC) ≥1000 cells/mm^3
  * Hemoglobin ≥12.0 g/dL for men and ≥11.0 g/dL for women
  * Platelet count ≥125,000/mm^3
  * Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m^2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) 2021 equation
  * Total bilirubin <1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (SGOT) <1.5 x ULN
  * Alanine aminotransferase (ALT) (SGPT) <1.5 x ULN
  * Alkaline phosphatase <1.5 x ULN
* Hepatitis C virus (HCV) antibody negative result within 60 days prior to Step 1 entry or, for participants who are HCV antibody positive (based on testing performed at any time prior to Step 1 entry), a negative HCV RNA result obtained within 60 days prior to Step 1 entry.
* Negative hepatitis B surface antigen (HBsAg) result obtained within 60 days prior to Step 1 entry.
* Ability and willingness to restart ART following ATI according to study guidelines.
* Completion of pre-entry leukapheresis or Large Volume Blood Draw (LVBD).

Exclusion Criteria:

* Breastfeeding or plans to become pregnant within the next 36 months.
* Known allergy/sensitivity or any hypersensitivity to components of study treatment or its formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Receipt of any investigational vaccine within 6 months prior to Step 1 entry.
* Receipt of any vaccine within 14 days prior to Step 1 entry.
* Prior receipt of anti-HIV broadly neutralizing antibody therapy.
* Prior receipt of a latency-reversing agent (LRA), whether licensed or investigational, unless reviewed and approved by the study's CMC.
* AIDS-defining illness or opportunistic infection within 24 months prior to Step 1 entry.
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases), other than HIV infection, that in the opinion of the investigator would preclude participation.
* Any history of an HIV-associated malignancy, including Kaposi's sarcoma and any type of lymphoma, or virus-associated cancers.
* History of progressive multifocal leukoencephalopathy (PML).
* Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery within 36 months prior to Step 1 entry or for whom such therapies are expected in the subsequent 12 months.
* Receipt of cabotegravir-LA intramuscular (IM) or rilpivirine-LA IM or lenacapavir (SQ) within 24 months prior to Step 1 entry.
* Resistance to one or more drugs in two or more ARV drug classes.
* History of systemic corticosteroids (long-term use), immunosuppressive anti-cancer or other immunosuppressive agents, interleukins, systemic interferons, systemic chemotherapy, or other medications considered significant by the investigator within the 6 months prior to Step 1 entry.
* History of or current clinical atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 ACC/AHA guidelines, including a previous diagnosis of any of the following:

  * Acute myocardial infarction
  * Acute coronary syndromes
  * Stable or unstable angina
  * Coronary or other arterial revascularization
  * Stroke
  * Transient ischemic attack
  * Peripheral arterial disease presumed to be of atherosclerotic origin
* For participants aged ≥40: 10-year ASCVD risk score estimated by Pooled Cohort Equations >20% within 60 days prior to Step 1 entry.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 60 days prior to Step 1 entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-08-29 (Estimated); Study Completion 2028-05-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing a Grade ≥3 Adverse Event (AE) or Serious Adverse Events (SAE) that are related to VRC07-523LS or PGT121.414.LS | Baseline through 36 weeks after the last dose of study treatment received
Proportion of study participants experiencing viral suppression, defined as HIV-1 RNA <200 copies/mL and remaining off ART | At 62 weeks after Step 1 entry

SECONDARY OUTCOMES:
Change from Step 1 entry in cell-associated HIV-1 RNA/DNA ratio in total CD4+ cells | Study entry through 72 weeks
  To be measured focusing on unspliced and single spliced env mRNA and corresponding total and env DNA.
Change from Step 1 entry in low-level viremia measured by single copy assay (SCA) | Study entry through 72 weeks
Change from Step 1 entry in levels of intact proviral DNA in CD4+ T-cells | Study entry through 72 weeks
Change from Step 1 entry in levels of inducible infectious virus on CD4+ T-cells | Study entry through 72 weeks
Average number of weeks from ATI until meeting the virologic criteria for ART restart | Week 2 through Week 72
Proportion of participants with HIV-1 RNA<1000 copies/mL | At 62 weeks
Serum concentrations of VRC07-523LS and PGT121.414.LS at the time meeting the virologic criteria for ART restart | At week 72
Area Under the Curve (AUC) of VRC07-523LS and PGT121.414.LS | Week 0 through End of Study, an average of 98 weeks
IC50 for neutralization sensitivity of the HIV-1 envelope population to VRC07-523LS and PGT121.414.LS | Week 0 through Week 72
Proportion of participants who develop antibodies to VRC07-523LS and PGT121.414.LS | Week 0 through End of Study, an average of 98 weeks
CD4+ T-cells counts | Week 0 through End of Study, an average of 98 weeks
HIV-1-specific T-cell count measured by Intracellular Cytokine Staining | Week 0 through Week 72

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Alabama CRS, Birmingham, Alabama
  - UCSD Antiviral Research Center CRS, San Diego, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - Houston Advancing Research Team CRS, Houston, Texas
- Brazil (2):
  - Instituto de Pesquisas em AIDS do Rio Grande do Sul - IPARGS CRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- Barranco CRS, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections) by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://submit.mis.s-3.net/
  Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.